CLINICAL TRIAL: NCT02828072
Title: Effects of Sudarshan Kriya Yoga on Cardiac Autonomic Control and Anxiety/Depression Levels in Patients Affected by Anxiety-Depression Disorders
Brief Title: Sudarshan Kriya Yoga and Cardiac Autonomic Control in Patients With Anxiety-Depression Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Eleonora Tobaldini, Doctor, University of Milan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKY-1
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sky (Experimental): Sky treatment foe 15 days
  Interventions: Other: SKY therapy
- control (Sham Comparator): standard medical therapy
  Interventions: Drug: usual drug therapy

INTERVENTIONS:
Other: SKY therapy — slow breathing
  Arms: Sky
Drug: usual drug therapy
  Arms: control

SUMMARY:
The effects of Sudarshan Kriya Yoga (SKY) on autonomic function in patients with anxiety-depression disorders is unknown. Thus, the authors will investigate cardiac autonomic control in a population of patients with anxiety-depression disorders which will undergo a specific SKY treatment.

DETAILED DESCRIPTION:
Several studies have demonstrated that adjuvant therapies as exercise and breathing training are effective in improving cardiac autonomic control (CAC) in patients with affective spectrum disorders. However, the effects of Sudarshan Kriya Yoga (SKY) on autonomic function in this population is unknown. To test the hypothesis that SKY training improves CAC, cardiorespiratory coupling and adaptive response of sympatho-vagal balance to orthostatic changes were evaluated in patients with anxiety and/or depression disorders.

The authors will enroll patients with a diagnosis of anxiety and/or depression disorders (DSM-IV) and they will divide them in two groups: 1) conventional therapy (Control) and 2) conventional therapy associated with SKY (Treatment) for 15 days. Anxiety and depression levels will be determined using quantitative questionnaires. For the assessment of CAC and cardiorespiratory coupling, cardiorespiratory traces will be analyzed using monovariate and bivariate autoregressive spectral analysis, respectively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of anxiety-depression disorder

Exclusion Criteria:

* absence of sinus rhythm on ECG
* absence of any cardiovascular and metabolic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in autonomic control | 1 month
  Parameter derived from heart rate variability: LF/HF (marker of sympatho-vagal balance)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toschi-Dias E, Tobaldini E, Solbiati M, Costantino G, Sanlorenzo R, Doria S, Irtelli F, Mencacci C, Montano N. Sudarshan Kriya Yoga improves cardiac autonomic control in patients with anxiety-depression disorders. J Affect Disord. 2017 May;214:74-80. doi: 10.1016/j.jad.2017.03.017. Epub 2017 Mar 7. PMID 28285240